CLINICAL TRIAL: NCT06805305
Title: Randomized Study of DOC1021 Dendritic Cell Immunotherapy in Combination With Standard of Care for Newly Diagnosed Adult Glioblastoma
Brief Title: DOC1021 Dendritic Cell Immunotherapy for Treatment of Newly Diagnosed Adult Glioblastoma (GBM)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Diakonos Oncology Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DOC-GBM2
Record Dates: First submitted 2025-01-14; First posted 2025-02-03 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Glioblastoma (GBM)
Keywords: Dendritic Cell Vaccine; Immunotherapy; Tumor vaccine
MeSH Terms: conditions — Glioblastoma | interventions — Transurethral Resection of Bladder; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DOC1021 + pIFN + SOC (Experimental): DOC1021 administered by injection near deep-cervical lymph nodes + pIFN adjuvant with standard of care treatment
  Interventions: Biological: DOC1021; Procedure: Tumor resection; Drug: Temodar (Temozolomide); Radiation: SOC cranial radiation
- SOC (Active Comparator): Standard of Care treatment alone
  Interventions: Procedure: Tumor resection; Drug: Temodar (Temozolomide); Radiation: SOC cranial radiation

INTERVENTIONS:
Biological: DOC1021 — Double-loaded dendritic cell vaccine, loaded with tumor lysate and mRNA using proprietary method
  Arms: DOC1021 + pIFN + SOC
Procedure: Tumor resection — SOC brain tumor resection
Drug: Temodar (Temozolomide) — SOC concomitant temozolomide during radiation and adjuvant temozolomide after radiation
Radiation: SOC cranial radiation — 60Gy radiation over 6 weeks in 2Gy fractions

SUMMARY:
The goal of this clinical trial is to learn if DOC1021 + pIFN alongside standard of care (SOC) will improve survival in adult patients newly diagnosed with glioblastoma (IDH-wt). It will also evaluate the safety of DOC1021 + pIFN. Researchers will compare DOC1021 dendritic cell immunotherapy regimen added to SOC compared to SOC treatment alone.

Participants in the DOC1021 + pIFN + SOC arm will:

* Take filgrastim subcutaneously x 5 doses and subsequently undergo a leukapheresis collection
* Undergo ultrasound guided perinodal DOC1021 injections every 2 weeks for a total of 3 doses
* Receive subcutaneous pIFN injections weekly for a total of 6 doses in parallel with the DOC1021 injections

Both arms of the trial will:

- Visit the clinic regularly to assess quality of life, symptoms, medication use, imaging, bloodwork, and to receive SOC treatment with surgery, temozolomide chemotherapy and radiation

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Age 18 years or older
4. Presumed diagnosis of glioblastoma IDH-wt (as per the 2021 WHO Classification of CNS Tumors) deemed to be potentially resectable and deemed to be a good candidate for post-operative standard of care temozolomide and radiation therapy.

   1. Surgical objective is for gross total resection (GTR)/near-total resection (NTR) de-fined as ≥ 95% of contrast enhancing (CE) tumor removed plus ≤ 1 cm3 residual CE tumor. Patients with subtotal resection will still be eligible if at least 70% of the CE tumor is resected.
   2. Eligibility will be confirmed after surgery when diagnosis of glioblastoma IDH-wt confirmed prior to randomization. Randomization can occur with only IDH1 immunohistochemistry and when additional molecular testing is available, if glioblastoma IDH-wt is not confirmed, the participant will be deemed a screen failure and replaced.
   3. Patients with prior biopsy or subtotal resection are eligible if no other anti-cancer treatment received for glioblastoma and additional resection indicated.
5. Ability to receive filgrastim (e.g., Neupogen), leukapheresis and 3 bi-weekly injections of DOC1021 near deep cervical lymph nodes + weekly pIFN x 6 weeks.
6. Females of reproductive potential must have a negative serum pregnancy test and agree to use effective contraception (as determined appropriate for the patient by the investigator) during study treatment.
7. Adequate kidney, liver, bone marrow function, and immune function, as follows:

   1. Hemoglobin ≥ 8.0 gm/dL
   2. Absolute neutrophil count (ANC) ≥ 1,500 cells/mm3
   3. Platelet count ≥ 75,000/mm3
   4. Calculated creatinine clearance (CrCl) > 30 mL/min using Cockcroft and Gault for-mula:

   i. For males = (140 - age[years]) x (body weight [kg]) / (72 x serum creatinine [mg/dL]) ii. For females = 0.85 x value from male formula e. Total bilirubin ≤ 1.5 times upper limit of normal (ULN) except in patients with Gilbert's disease for which total bilirubin must be ≤ 2 times ULN f. Aspartate transaminase AST (SGOT) and alanine aminotransferase ALT (SGPT) ≤ 3 times the ULN
8. Karnofsky Performance Score ≥ 70

Exclusion Criteria:

1. Infratentorial, recurrent, leptomeningeal or extracranial disease.
2. Patients who are pregnant or breastfeeding.
3. Known active HIV or hepatitis infection. Patients with HIV that is well-controlled and have undetectable viral titers remain eligible. Patients with history of HCV adequately treated such that RNA viral load is negative also remain eligible.
4. Any severe or uncontrolled medical condition or other condition that could affect participation in this study as determined by the investigator, including but not limited to: uncontrolled or severe cardiac disease, systemic autoimmune disorders requiring immunosuppression in the past 2 years*, autoimmune hyper/hypothyroidism, untreated viral hepatitis, autoimmune hepatitis. *autoimmune disorders include but are not limited to rheumatoid arthritis, psoriasis and inflammatory bowel disease and immunosuppressive medications include DMARDs like methotrexate, TNF inhibitors, IL-6 receptor blockers, CD80/86 inhibitors, anti-CD20 and JAK inhibitors
5. Treatment with another investigational drug or other experimental intervention within the last 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2030-03 (Estimated); Study Completion 2032-03 (Estimated)

PRIMARY OUTCOMES:
Overall survival (time in months from randomization until death for each participant) | 5 years

SECONDARY OUTCOMES:
Number of total participants treated with DOC1021 alive at one year post-GBM diagnosis date | 1 years
  One-year survival
Number of total participants treated with DOC1021 alive two years post-GBM diagnosis date | 2 years
  2-year survival rate
Number of total participants treated with DOC1021 alive three years post-GBM diagnosis date | 3 years
  3-year survival
Number of Participants with Adverse Events as Assessed by CTCAE v5.0 | 3 years
Time in months from initial diagnosis of new diagnosed GBM until declared progression on imaging by RANO 2.0 criteria for all participants | 3 years

OTHER OUTCOMES:
Health-related quality of life in all participants as assessed by EORTC Quality of Life Questionnaire Cancer QLC-C30 (Cancer 30-items) with QLQ-BN20 (Brain 20-items) module included. | 5 years
  All items are scored 1 (worse outcome) to 4 (better outcome) or 1 (worse outcome) to 7 (better outcome). All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Neuro-cognitive function in all participants as Assessed by the Neurologic Assessment in Neuro-Oncology (NANO) scale | 5 years

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - City of Hope, Duarte, California
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Rutgers Cancer Institute, New Brunswick, New Jersey
  - Atlantic Health, Summit, New Jersey
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania
  - UTHealth Houston, Houston, Texas
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No